CLINICAL TRIAL: NCT04467944
Title: Effect of Pre-existing Adjacent Segment Degeneration on Long-term Effectiveness After Lumbar Fusion Surgery: a Prospective Cohort Study
Brief Title: Effect of Pre-existing Adjacent Segment Degeneration on Long-term Effectiveness After Lumbar Fusion Surgery
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2017399
Record Dates: First submitted 2020-06-28; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-06

CONDITIONS: Degenerative Lumbar Spinal Stenosis; Degenerative Disc Disease; Degeneration Spine
Keywords: Cerebrospinal fluid occlusion; Pre-existing degeneration; Spinal canal stenosis; Adjacent segment degeneration; Adjacent segment disease; High-intensity zone; Vacuum sign
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NS Group: Patients without pre-existing degeneration at L3/4 segment will be classified into control group (NS group).
- D Group: Patients with pre-existing disc factors (Pfirrmann grade≥3, Hiz or vacuum sign) at L3/4 segment will be classified into group D.
  Interventions: Other: Pre-existing degenerative factors at adjacent segment
- C Group: Patients with pre-existing canal stenosis factors (cerebrospinal fluid occlusion≥1) at L3/4 segment will be classified into group C.
  Interventions: Other: Pre-existing degenerative factors at adjacent segment

INTERVENTIONS:
Other: Pre-existing degenerative factors at adjacent segment — Pre-existing degenerative factors at adjacent segment, including disc factors and canal stenosis factors
  Groups: C Group; D Group

SUMMARY:
This is a prospective single-center study. Patients requiring posterior lumbar interbody fusion (PLIF) for lumbar degenerative disease are prospectively enrolled and followed. Important adjacent pre-existing degeneration factors include discs degenerated, facets and ligamentum flavum tropism which could lead to spinal canal stenosis (SCS). This study will focus on the effects of pre- existing adjacent degeneration (disc factors and spinal canal stenosis factors) on long-term postoperative outcomes.

DETAILED DESCRIPTION:
Adjacent segment pathologies (ASP), including radiological adjacent segment degeneration (ASDeg) and adjacent segment disease (ASDis) after lumbar fusion surgeries have been troubling complications. The development of ASDis greatly reduces postoperative quality of life, and revision surgery may be required in severe cases. Several risk factors for ASP have been reported, such as age, sex, pre-existing adjacent degeneration, multilevel fusions, sagittal imbalance, the type of fusion, facet tropism and laminar inclination. Because multi-level degenerative imaging is common in lumbar degenerative disease, pre-existing adjacent degeneration makes challenge for the surgery strategy, sometimes it is difficult to determine the level at which fusion ends. Important pre-existing adjacent degeneration factors included discs degenerated, facets and ligamentum flavum tropism which could lead to spinal canal stenosis (SCS). Few studies have focused on asymptomatic pre-existing SCS as a risk factor for ASDis that requires additional surgery at an adjacent segment. But these studies only used the sagittal diameter or ratio to evaluate the degree of adjacent SCS. The status of neural tissues in the canal was neglected. Few studies also have focused on asymptomatic pre-existing degenerated disc as a risk factor for ASDeg. But these studies only used Pfirrmann grade to evaluate the degenerated disc. High-intensity zone (Hiz), vacuum sign were neglected.

This prospective study was limited to patients with the same preoperative pathology, the same fusion segments (L4-5 and L5-S1), the same fusion technique (PLIF). Dynamic X-ray and MRI examinations of lumbar will be completed to evaluate the imaging manifestations of the responsible and adjacent segments before surgery. The T2-weighted sagittal and axial MRI images are studied and the following parameters are recorded: grade of cerebrospinal fluid occlusion in L3/4 spinal canal at disc level, and the narrowest axial plane was used for grading; L3/4 disc degeneration by Pfirrmann grade; high-intensity zone (Hiz) and vacuum sign of L3/4 disc; L3/4 disc herniation quantificationally measured by MSU Classification; Patients will be divided into three groups according to the pre-existing status of L3/4 segment. Patients without pre-existing degeneration at L3/4 segment will be classified into control group (NS group). Patients with pre-existing disc factors (Pfirrmann grade≥3, Hiz or vacuum sign) at L3/4 segment will be classified into group D. Patients with pre-existing canal stenosis factors (cerebrospinal fluid occlusion≥1) at L3/4 segment will be classified into group C.

The patient's age, gender, preoperative body mass index (BMI), American Society of Anesthesiologists classification of anesthesia (ASA grade) will be recorded during the hospital stay. Surgical data including operation time, blood loss, perioperative complications (including cerebrospinal fluid leakage, wound infection, postoperative neurological dysfunction, and perioperative secondary surgery, cardiopulmonary complication, cerebral infarction/hemorrhage, etc.), and length of hospital stay are also recorded. Preoperative clinical function questionnaires, including visual analog scale (VAS) of low back, VAS of the legs, and Oswestry Disability Index (ODI) scores for patients were completed on admission for surgery without any assistance. All the patients enrolled will finished the follow-up from date of surgery at 1,2 and 5 years. The clinical outcomes and ASP will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* A clear diagnosis of lumbar spinal stenosis, and surgical level of L4- S1 (The levels to be operated on were decided by matching the clinical symptomatology with the radiological findings of the spinal levels that needed decompression);
* Failed at least eight weeks conservative treatment;

Exclusion Criteria:

* Unstable factors (slip, rotation, lateral bending, etc.) in adjacent segment L3/4;
* Preoperative sagittal and coronal imbalance of the spine;
* Lumbar infection and/or tumor diseases;
* A previous history of lumbar fusion surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the orthopaedic department of Peking University Third Hospital, patients with a clear diagnosis of lumbar degenerative disease, and surgical level of L4-S1 will be enrolled.
Sampling Method: Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Adjacent segment degeneration (ASDeg) | 12 months after surgery
  ASDeg is defined as follows according to manifestations on X-rays and MRI changing from baseline : (1) Progression ≥1 grade in SCS or L3/4 disc degeneration; (2)Alteration of L3/4 disc herniation, Hiz and vacuum sign; (3) Progression of ≥ 3 mm in vertebral slippage, a change of ≥ 10° in the intervertebral angle on flexion and extension lateral radiograph, or scoliosis deformity on coronal plane.
Adjacent segment degeneration (ASDeg) | 24 months after surgery
  ASDeg is defined as follows according to manifestations on X-rays and MRI changing from baseline : (1) Progression ≥1 grade in SCS or L3/4 disc degeneration; (2)Alteration of L3/4 disc herniation, Hiz and vacuum sign; (3) Progression of ≥ 3 mm in vertebral slippage, a change of ≥ 10° in the intervertebral angle on flexion and extension lateral radiograph, or scoliosis deformity on coronal plane.
Adjacent segment degeneration (ASDeg) | 60 months after surgery
  ASDeg is defined as follows according to manifestations on X-rays and MRI changing from baseline : (1) Progression ≥1 grade in SCS or L3/4 disc degeneration; (2)Alteration of L3/4 disc herniation, Hiz and vacuum sign; (3) Progression of ≥ 3 mm in vertebral slippage, a change of ≥ 10° in the intervertebral angle on flexion and extension lateral radiograph, or scoliosis deformity on coronal plane.
Adjacent segment degeneration (ASDeg) | 120 months after surgery
  ASDeg is defined as follows according to manifestations on X-rays and MRI changing from baseline : (1) Progression ≥1 grade in SCS or L3/4 disc degeneration; (2)Alteration of L3/4 disc herniation, Hiz and vacuum sign; (3) Progression of ≥ 3 mm in vertebral slippage, a change of ≥ 10° in the intervertebral angle on flexion and extension lateral radiograph, or scoliosis deformity on coronal plane.
Adjacent segment disease (ASDis) | The entire study process, up to 120 months after surgery.
  ASDis is defined as clinical and radiographic evidence of degenerative spinal disease (disc degeneration, stenosis, or spondylolisthesis) on the level adjacent to the index fusion.

SECONDARY OUTCOMES:
Disability | 12 months after surgery; 24 months after surgery; 60 months after surgery; 120 months after surgery.
  The Oswestry Disability Index (ODI) (0-100) is used to assess disability.
Back pain | 12 months after surgery; 24 months after surgery; 60 months after surgery; 120 months after surgery.
  The Visual Analog Scale (0-10) is used to evaluate back pain.
Leg pain | 12 months after surgery; 24 months after surgery; 60 months after surgery; 120 months after surgery.
  The Visual Analog Scale (0-10) is used to evaluate leg pain.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Shi Li, Dr., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
We will make the clinical study report available for half a year after the publication of the results of the study.
Supporting Information: CSR
Time Frame: The IPD will become available for half a year after the publication of the results of the study.
Access Criteria: The IPD is available to the readers of the journal in which our research is published. The corresponding author of the published papers will review the requests.

REFERENCES:
- [Result] Lee JC, Kim Y, Soh JW, Shin BJ. Risk factors of adjacent segment disease requiring surgery after lumbar spinal fusion: comparison of posterior lumbar interbody fusion and posterolateral fusion. Spine (Phila Pa 1976). 2014 Mar 1;39(5):E339-45. doi: 10.1097/BRS.0000000000000164. PMID 24365899
- [Result] Lawrence BD, Wang J, Arnold PM, Hermsmeyer J, Norvell DC, Brodke DS. Predicting the risk of adjacent segment pathology after lumbar fusion: a systematic review. Spine (Phila Pa 1976). 2012 Oct 15;37(22 Suppl):S123-32. doi: 10.1097/BRS.0b013e31826d60d8. PMID 22885827
- [Result] Yugue I, Okada S, Masuda M, Ueta T, Maeda T, Shiba K. Risk factors for adjacent segment pathology requiring additional surgery after single-level spinal fusion: impact of pre-existing spinal stenosis demonstrated by preoperative myelography. Eur Spine J. 2016 May;25(5):1542-1549. doi: 10.1007/s00586-015-4185-6. Epub 2015 Aug 14. PMID 26272373
- [Result] Lee GY, Lee JW, Choi HS, Oh KJ, Kang HS. A new grading system of lumbar central canal stenosis on MRI: an easy and reliable method. Skeletal Radiol. 2011 Aug;40(8):1033-9. doi: 10.1007/s00256-011-1102-x. Epub 2011 Feb 1. PMID 21286714
- [Result] Mysliwiec LW, Cholewicki J, Winkelpleck MD, Eis GP. MSU classification for herniated lumbar discs on MRI: toward developing objective criteria for surgical selection. Eur Spine J. 2010 Jul;19(7):1087-93. doi: 10.1007/s00586-009-1274-4. Epub 2010 Jan 19. PMID 20084410
- [Result] Nakashima H, Kawakami N, Tsuji T, Ohara T, Suzuki Y, Saito T, Nohara A, Tauchi R, Ohta K, Hamajima N, Imagama S. Adjacent Segment Disease After Posterior Lumbar Interbody Fusion: Based on Cases With a Minimum of 10 Years of Follow-up. Spine (Phila Pa 1976). 2015 Jul 15;40(14):E831-41. doi: 10.1097/BRS.0000000000000917. PMID 25839385